CLINICAL TRIAL: NCT00548405
Title: A Phase 3, Randomized, Rater- and Dose-Blinded Study Comparing Two Annual Cycles of Intravenous Low- and High-Dose Alemtuzumab to Three-Times Weekly Subcutaneous Interferon Beta 1a (Rebif®) in Patients With Relapsing Remitting Multiple Sclerosis Who Have Relapsed On Therapy
Brief Title: Comparison of Alemtuzumab and Rebif® Efficacy in Multiple Sclerosis, Study Two
Acronym: CARE-MS II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAMMS32400507; 2007-001162-32 (EudraCT Number); CAMMS324,; ISRCTN70702834 (Registry Identifier: ISRCTN); ACTRN12608000426381 (Registry Identifier: ANZCTR); NTR1469 (Registry Identifier: The Netherlands National Trial Register); CARE-MS II (Other: NMSS)
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Alemtuzumab; Interferon beta-1a

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alemtuzumab 12 mg (Experimental): Alemtuzumab (Lemtrada™) 12 milligram (mg) per day intravenous (IV) infusion on 5 consecutive days at Month 0, followed by alemtuzumab 12 mg per day IV infusion on 3 consecutive days at Month 12.
  Interventions: Biological: Alemtuzumab 12 mg
- Alemtuzumab 24 mg (Experimental): Alemtuzumab 24 mg per day IV infusion on 5 consecutive days at Month 0, followed by alemtuzumab 24 mg per day IV infusion on 3 consecutive days at Month 12.
  Interventions: Biological: Alemtuzumab 24 mg
- Interferon Beta-1a (Active Comparator): Interferon Beta-1a (Rebif®) 44 microgram (mcg) subcutaneously 3-times weekly for 24 months. Dose adjustment was done as per Investigator's discretion.
  Interventions: Biological: Interferon beta-1a

INTERVENTIONS:
Biological: Alemtuzumab 12 mg — Alemtuzumab 12 milligram (mg) per day intravenous (IV) infusion on 5 consecutive days at Month 0, followed by alemtuzumab 12 mg per day IV infusion on 3 consecutive days at Month 12.
  Other Names: Lemtrada
  Arms: Alemtuzumab 12 mg
Biological: Alemtuzumab 24 mg — Alemtuzumab 24 mg per day IV infusion on 5 consecutive days at Month 0, followed by alemtuzumab 24 mg per day IV infusion on 3 consecutive days at Month 12.
  Other Names: Lemtrada
  Arms: Alemtuzumab 24 mg
Biological: Interferon beta-1a — Interferon beta-1a 44 microgram (mcg) subcutaneously 3-times weekly for 24 months. Dose adjustment was done as per Investigator's discretion.
  Other Names: Rebif®
  Arms: Interferon Beta-1a

SUMMARY:
The purpose of this study was to establish the efficacy and safety of two different doses of alemtuzumab (Lemtrada™) as a treatment for relapsing-remitting multiple sclerosis (MS), in comparison with subcutaneous interferon beta-1a (Rebif®). The study enrolled participants who had received an adequate trial of disease-modifying therapies but experienced at least 1 relapse during prior treatment, and who met a minimum severity of disease as measured by magnetic resonance imaging (MRI). Participants had monthly laboratory tests and comprehensive testing every 3 months.

DETAILED DESCRIPTION:
Every participant received active treatment; there was no placebo. After Amendment 2, the 24 mg alemtuzumab dose was closed to enrollment so newly enrolled participants were randomly assigned to treatment with either 12 mg alemtuzumab or interferon beta-1a in a 2:1 ratio (that is, 2 given 12 mg alemtuzumab for every 1 given interferon beta-1a). Alemtuzumab was administered in two annual courses, once at the beginning of the study and again 1 year later. Interferon beta-1a was self-injected 3 times per week for 2 years. All participants were required to return to their study site every 3 months for neurologic assessment. In addition, safety-related laboratory tests were performed at least monthly. Participation in this study ended 2 years after the start of treatment for each participant. Additionally, participants who received alemtuzumab might be followed in the CAMMS03409 Extension Study (NCT00930553) for safety and efficacy assessments. Participants who received interferon beta-1a and completed 2 years on study might be eligible to receive alemtuzumab in the Extension Study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF)
* Age 18 to 55 years (inclusive) as of the date the ICF was signed
* Diagnosis of MS per update of McDonald criteria
* Onset of MS symptoms (as determined by a neurologist; could be retrospectively) within 10 years of the date the ICF was signed
* Expanded Disability Status Scale (EDSS) score 0.0 to 5.0 (inclusive) at Screening
* Greater than or equal to (>=) 2 MS attacks (first episode or relapse) occurring in the 24 months prior to the date the ICF was signed, with >=1 attack in the 12 months prior to the date the ICF was signed, with objective neurological signs confirmed by a physician, nurse practitioner, or other Genzyme-approved health-care provider and the objective signs could be identified retrospectively
* >=1 MS relapse during treatment with a beta interferon therapy or glatiramer acetate after having been on that therapy for >=6 months within 10 years of the date the ICF was signed
* MRI scan demonstrating white matter lesions attributable to MS and meeting at least 1 of the following criteria, as determined by the neurologist or a radiologist: >=9 time constant 2 (T2) lesions at least 3 millimeter (mm) in any axis; a gadolinium- (Gd-) enhancing lesion at least 3 mm in any axis plus >=1 brain T2 lesions; and a spinal cord lesion consistent with MS plus >=1 brain T2 lesion

Exclusion Criteria:

* Received prior therapy with alemtuzumab
* Current participation in another clinical study or previous participation in CAMMS323 (Comparison of Alemtuzumab and Rebif Efficacy in Multiple Sclerosis, CARE-MS I)
* Treatment with natalizumab, methotrexate, azathioprine, or cyclosporine in the past 6 months. Participants who received one of these medications more than 6 months before the date the ICF was signed were eligible for study entry if approval was granted by Genzyme
* Any progressive form of MS
* History of malignancy (except basal skin cell carcinoma)
* CD4 +, CD8 +, CD19 + (that is, absolute CD3 + CD4 + , CD3 + CD8 + , or CD19 + /mm 3 ) count, absolute neutrophil count less than (<) lower limit of normal (LLN) at screening; if abnormal cell count(s) returned to within normal limits (WNL), eligibility could be reassessed
* Known bleeding disorder (for example, dysfibrinogenemia, factor IX deficiency, hemophilia, Von Willebrand's disease, disseminated intravascular coagulation, fibrinogen deficiency, or clotting factor deficiency)
* Significant autoimmune disease including but not limited to immune cytopenias, rheumatoid arthritis, systemic lupus erythematosus, other connective tissue disorders, vasculitis, inflammatory bowel disease, severe psoriasis
* Presence of anti-thyroid stimulating hormone (TSH) receptor (TSHR) antibodies (that is, above the LLN)
* Active infection or at high risk for infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 840 (Actual)
Dates: Start 2007-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (191):
- United States (85):
  - North Central Neurology Associates, P.C., Cullman, Alabama
  - Barrow Neurological Institute, St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - Mayo Clinic Arizona, Department of Neurology, Scottsdale, Arizona
  - Northwest NeuroSpecialists, PLLC, Tucson, Arizona
  - East Bay Physicians Medical Group/Sutter East Bay Medical Foundation, Berkeley, California
  - Neurology Center of North Orange County, La Habra, California
  - Department of Neurology, Keck School of Medicine, University of Southern California, Los Angeles, California
  - Neuro-Therapeutics Inc., Pasadena, California
  - Neuro-Therapeutics, Inc, Pasadena, California
  - University of California, Davis Medical Center, Sacramento, California
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado Hospital, Anschutz Outpatient Pavilioin, Aurora, Colorado
  - Neurological Consultants, Denver, Colorado
  - Advanced Neurosciences Research, Fort Collins, Colorado
  - Yale University, New Haven, Connecticut
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - University of Florida Neuroscience Institute, Jacksonville, Florida
  - Neurology Associates, P.A., Maitland, Florida
  - Neurological Associates, Pompano Beach, Florida
  - Negroski, Stein, Sutherland and Hanes Neurology, Sarasota, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - University of South Florida, Department of Neurology, Tampa, Florida
  - Emory University, Department of Neurology, Atlanta, Georgia
  - Shepherd Center, Inc., Atlanta, Georgia
  - Idaho Falls Multiple Sclerosis Center, PLLC, Idaho Falls, Idaho
  - University of Chicago Medical Center, Department of Neurology, Chicago, Illinois
  - Consultants in Neurology, Ltd, Northbrook, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Indiana University School of Medicine, Department of Neurology, Indianapolis, Indiana
  - Josephson Wallack Munshower Neurology P.C., Indianapolis, Indiana
  - Iowa Health Physicians, Des Moines, Iowa
  - Ruan Neurology Clinic and Research Center, Des Moines, Iowa
  - University of Kansas Medical Center, Department of Neurology, Kansas City, Kansas
  - MidAmerica Neuroscience Institute, Lenexa, Kansas
  - Associates in Neurology, PSC, Lexington, Kentucky
  - University of Louisville Research Foundation, Louisville, Kentucky
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Partners Multiple Sclerosis Center/Brigham and Women's Hospital, Boston, Massachusetts
  - Springfield Neurology Associates, LLC, Springfield, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Department of Neurology, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Wayne State University, School of Medicine, Department of Neurology, Detroit, Michigan
  - Spectrum Health Medical Group, Neurology (Previously known as Michigan Medical P.C., Neurology), Grand Rapids, Michigan
  - Michigan Neurology Associates, P.C., Saint Clair Shores, Michigan
  - Northern Michigan Neurology, Traverse City, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Neurology Consultants of Kansas City, Inc., Kansas City, Missouri
  - Montana Neurobehavioral Specialists, Missoula, Montana
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Renown Institute for Neurosciences / Renown regional Medical Center, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center, Norris Cotton Cancer Center, Lebanon, New Hampshire
  - MS Center at Holy Name Hospital, Teaneck, New Jersey
  - University of New Mexico, Health Sciences Center, MS Specialty Clinic, Albuquerque, New Mexico
  - Empire Neurology, PC, Latham, New York
  - Winthrop University Hospital, Clinical Trials Center, Mineola, New York
  - Mount Sinai School of Medicine, Corinne Goldsmith Dickinson Center for Multiple Sclerosis, New York, New York
  - Comprehensive Multiple Sclerosis Care Center at South Shore Neurologic Associates, P.C., Patchogue, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Department of Neurology, Syracuse, New York
  - University of North Carolina-Chapel Hill, Department of Neurology, Chapel Hill, North Carolina
  - Wake Forest University Health Science, Department of Neurology, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Mellen Center, Cleveland, Ohio
  - Neurology Specialists, Inc., Dayton, Ohio
  - Oak Clinic for Multiple Sclerosis, Uniontown, Ohio
  - MS Center of Oklahoma, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital, Neuroscience and Pain Research, Allentown, Pennsylvania
  - Northshore Clinical Associates, Erie, Pennsylvania
  - University of Pittsburgh, Kaufmann Medical Building, Pittsburgh, Pennsylvania
  - The Neurology Foundation, Inc., Providence, Rhode Island
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Advanced Neurosciences Institute, Franklin, Tennessee
  - Biomedical Research Alliance of NY, LLC, Franklin, Tennessee
  - Hope Neurology PC, Knoxville, Tennessee
  - Vanderbilt Multiple Sclerosis Center, Nashville, Tennessee
  - Clinical Center for Multiple Sclerosis, Dallas, Texas
  - Central Texas Neurology, Round Rock, Texas
  - Integra Clinical Research, San Antonio, Texas
  - Neurology Center of San Antonio, San Antonio, Texas
  - MS Center of Greater Washington, P.C., Vienna, Virginia
  - Swedish Neuroscience Institute, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Rockwood Clinical Research Center, Spokane, Washington
- DIABAID, Buenos Aires, Argentina
- Australia (11):
  - Westmead Hospital, Westmead, New South Wales
  - The Wesley Research Institute, Auchenflower, Queensland
  - Griffith School of Medicine, Gold Coast Campus, Griffith University, Southport, Queensland
  - Clinical Cognitive Research Unit/Clinical Trials, The Queen Elizabeth Hospital, Neurology Department, Woodville South, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - St. Vincent's Hospital, MS Education & Research, Department of Clinical Neurosciences, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Department of Neurology, Parkville, Victoria
  - Concord Repatriation General Hospital, Neurosciences Department, Concord
  - Southern Neurology, Kogarah
  - Liverpool Hospital, Neurology Department, Liverpool
- AKH Wien, Universitätsklinikum für Neurologie, Vienna, Austria
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Neurology, Brussels
  - CHU Ourthe Amblève, Neurology, Esneux
  - University Hospital Leuven, Campus Gasthuisberg, Neurology, Leuven
- Brazil (4):
  - Hospital da Restauracao, Recife, Pernambuco
  - Hospital Sao Lucas PUC-RS, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas USP, São Paulo
  - Irmandade da Santa Casa de Misericordia de Sao Paulo, São Paulo
- Canada (9):
  - UBC Hospital, Vancouver, British Columbia
  - Multiple Sclerosis Clinic, Connell 7, Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre- University Hospital, London, Ontario
  - The Ottawa Hospital, General Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre de Sante et de Services Sociaux de Gatineau-Hull Hospital, Gatineau, Quebec
  - Clinique Neuro rive-sud, Recherche sepmus inc, Greenfield Park, Quebec
  - Hospital Maisonneuve-Rosemont, Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- Croatia (5):
  - Clinical Hospital Centre Rijeka, Clinic for Neurology, Rijeka
  - General Hospital Varazdin, Department of neurology, Varaždin
  - Clinical Hospital Centre Zagreb, Zagreb
  - Clinical Hospital Sestre Milosrdnice, Zagreb
  - General Hospital " Sveti Duh", Department of neurology, Zagreb
- Czechia (4):
  - MS Center, Department of Neurology, Hradec Králové
  - St. Anne's University Hospital Brno, Pekarska
  - Department of Neurology 1st Faculty of Medicine and General Teaching Hospital, MS Center, Prague
  - Krajska zdravotni a.s. - Hospital Teplice, Teplice
- Denmark (3):
  - Århus Universitetshospital, Scleroseklinikken, Århus Sygehus, Aarhus
  - Scleroseklinikken, Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- France (6):
  - CHU Clermont-Ferrand, Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital General, Service de Neurologie, Dijon
  - Hospital Roger Salengro, Lille
  - Hôpital Pitié Salpétrière, Service de Neurologie, Paris
  - Sevice de Neurologie, Rennes
  - Hôpital Civil, Departement de Neurologie, Strasbourg
- Germany (13):
  - Krankenhaus Hohe Warte, Betriebsstätte der Bayreuth, Bayreuth
  - Judisches Krankenhaus Berlin, Berlin
  - Neurologisches Fachzentrum Berlin, Berlin
  - Neurologische Universitätsklinik Bonn, Bonn
  - Multiple Sklerose Zentrum am, Zentrum für klinische Neurowissenschaften, Neurologische Uniklinik Dresden, Dresden
  - Asklepios Klinic Barmbek, Hamburg
  - Medizinische Hochshule Hannover, Hanover
  - Oberhavelkliniken Hennigsdorf, Hennigsdorf
  - Klinikum Ingolstadt, Neurologische Klinik, Ingolstadt
  - Klinikum Rechts der Isar, Klinik für Neurologie, München
  - Klinik und Poliklinik fur Neurologie der Universitat Rockstock, Rostock
  - Universitatsklinik Ulm, Ulm
  - Fachkrankenhaus Hubertusburg, Wermsdorf
- Israel (3):
  - Hadassah Medical Center Ein Karem, Jerusalem
  - Tel Aviv Sourasky Medical Center, Department of Neurology, Tel Aviv
  - Sheba Medical Centre, Tel Litwinsky
- Italy (6):
  - Ospedale Binaghi - Centro Sclerosi Multipla, Cagliari
  - Ospedale S. Antonio Abate di Gallarate, Gallarate
  - Università di Genova Dipartimento di Neuroscienze Oftalmologia e Genetica, Genova
  - Ospedale Civile di Brescia c/o Ospedale Richiedei, Centro di riferimento per la Sclerosi Multiple, Montichiari
  - Ospedale San Luigi di Orbassano, Orbassano
  - Azienda Ospedaliera Sant'Andrea Neurologia, Roma
- Mexico (3):
  - Unidad de Investigación en Salud de Chihuahua, S.C., Chihuahua City, Chihuahua
  - Hospital Medica Sur CIF-BIOTEC, Delegacion, Tlalpan
  - Hospital Angeles del Pedregal; Camino a Santa Teresa, Mexico City
- Netherlands (2):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Orbis Medisch Centrum, Department of Neurology, Sittard
- Poland (3):
  - Independent Public Healthcare Facility, Norbert Barlicki University Hospital No. 1 of the Medical University of Lodz, Lodz
  - Independent Public Teaching Hospital No. 4 in Lublin, Lublin
  - Heliodor Swiecicki Teaching Hospital of the Poznan, University of Medical Sciences, Poznan
- Russia (11):
  - Research Medical Complex "Your Health" Ltd, Kazan'
  - Institution of the Russian Academy of Medical Sciences, "Neurology Scientific Center under RAMS", Moscow
  - Moscow State Medical Institution City Clinical Hospital #11, Moscow City Center for Multiple Sclerosis, Moscow
  - Moscow State Public Medical Institution, City Clinical Hospital #11, Moscow
  - Municipal Treatment and Prevention Institution, "City Hospital #33", Nizhny Novgorod
  - Federal State Institution: Siberian District Medical Center, Novosibirsk
  - Institution of the Russian Academy of Sciences, "Institute of the Human Brain n.a. N.P. Bekhtereva within the Russian Academy of Sciences", Saint Petersburg
  - St. Petersburg Pavlov State Medical University, Department of Neurology and Neurosurgery with a Clinic, Saint Petersburg
  - St.Petersburg State Medical Institution, "City Multispecialty Hospital #2", Saint Petersburg
  - St.Petersburg State Medical Institution, "Nikolayevskaya Hospital", Saint Petersburg
  - State Medical Institution, "Samara Regional Clinical Hospital n.a. M.I. Kalinin", Samara
- Serbia (4):
  - Clinic of Neurology, Clinical Centre of Serbia, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Centre of Kragujevac, Kragujevac
  - Clinical Centre Vojvodina Institute of Neurology, Novi Sad
- Spain (4):
  - Servicio de Neurología Hospital Vall d'Hebron Paseo de Vall d'Hebron, Barcelona
  - Servicio de Neurología Hospital Clínico San Carlos, Madrid
  - Servicio de Neurología Hospital Carlos Haya, Málaga
  - Servicio de Neurología Hospital Virgen de la Macarena, Seville
- Sweden (2):
  - Sahlgrenska University Hospital, Neurologkliniken, Gothenburg
  - Norrlands Universitets sjukhus, Umeå
- Ukraine (3):
  - Institute of Neurology, Psychiatry and Narcology under the Academy of Medical Sciences of Ukraine, Kharkiv
  - Kyiv Municipal Clinical Hospital #4, Department of Demyelinating Diseases of the Nervous System, Kyiv
  - Danylo Halytsky Lviv National Medical University, Department of Neurology, Lviv
- United Kingdom (5):
  - Department Of Neurosciences, Addenbrookes Hospital, Cambridge, England
  - Centre for Neuroscience & Trauma, Blizard Institute of Cell and Molecular Science Barts and The London School of Medicine and Dentistry, London, England
  - Frenchay Hospital, Bristol
  - Salford Royal NHS Foundation Trust, Clinical Trials Unit, Salford
  - Department of Neurology Glossop Road, Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Background] Coles AJ, Twyman CL, Arnold DL, Cohen JA, Confavreux C, Fox EJ, Hartung HP, Havrdova E, Selmaj KW, Weiner HL, Miller T, Fisher E, Sandbrink R, Lake SL, Margolin DH, Oyuela P, Panzara MA, Compston DA; CARE-MS II investigators. Alemtuzumab for patients with relapsing multiple sclerosis after disease-modifying therapy: a randomised controlled phase 3 trial. Lancet. 2012 Nov 24;380(9856):1829-39. doi: 10.1016/S0140-6736(12)61768-1. Epub 2012 Nov 1. PMID 23122650
- [Derived] Ziemssen T, Bass AD, Van Wijmeersch B, Eichau S, Richter S, Hoffmann F, Armstrong NM, Chirieac M, Cunha-Santos J, Singer BA. Long-term efficacy and safety of alemtuzumab in participants with highly active MS: TOPAZ clinical trial and interim analysis of TREAT-MS real-world study. Ther Adv Neurol Disord. 2025 Feb 10;18:17562864241306575. doi: 10.1177/17562864241306575. eCollection 2025. PMID 39935588
- [Derived] Coles AJ, Achiron A, Traboulsee A, Singer BA, Pozzilli C, Oreja-Guevara C, Giovannoni G, Comi G, Freedman MS, Ziemssen T, Shiota D, Rawlings AM, Wong AT, Chirieac M, Montalban X. Safety and efficacy with alemtuzumab over 13 years in relapsing-remitting multiple sclerosis: final results from the open-label TOPAZ study. Ther Adv Neurol Disord. 2023 Sep 21;16:17562864231194823. doi: 10.1177/17562864231194823. eCollection 2023. PMID 37745914
- [Derived] Riera R, Torloni MR, Martimbianco ALC, Pacheco RL. Alemtuzumab for multiple sclerosis. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD011203. doi: 10.1002/14651858.CD011203.pub3. PMID 37272540
- [Derived] Dayan CM, Lecumberri B, Muller I, Ganesananthan S, Hunter SF, Selmaj KW, Hartung HP, Havrdova EK, LaGanke CC, Ziemssen T, Van Wijmeersch B, Meuth SG, Margolin DH, Poole EM, Baker DP, Senior PA. Endocrine and multiple sclerosis outcomes in patients with autoimmune thyroid events in the alemtuzumab CARE-MS studies. Mult Scler J Exp Transl Clin. 2023 Jan 3;9(1):20552173221142741. doi: 10.1177/20552173221142741. eCollection 2023 Jan-Mar. PMID 36619856
- [Derived] Coles AJ, Jones JL, Vermersch P, Traboulsee A, Bass AD, Boster A, Chan A, Comi G, Fernandez O, Giovannoni G, Kubala Havrdova E, LaGanke C, Montalban X, Oreja-Guevara C, Piehl F, Wiendl H, Ziemssen T. Autoimmunity and long-term safety and efficacy of alemtuzumab for multiple sclerosis: Benefit/risk following review of trial and post-marketing data. Mult Scler. 2022 Apr;28(5):842-846. doi: 10.1177/13524585211061335. Epub 2021 Dec 9. PMID 34882037
- [Derived] Coles AJ, Arnold DL, Bass AD, Boster AL, Compston DAS, Fernandez O, Havrdova EK, Nakamura K, Traboulsee A, Ziemssen T, Jacobs A, Margolin DH, Huang X, Daizadeh N, Chirieac MC, Selmaj KW. Efficacy and safety of alemtuzumab over 6 years: final results of the 4-year CARE-MS extension trial. Ther Adv Neurol Disord. 2021 Apr 23;14:1756286420982134. doi: 10.1177/1756286420982134. eCollection 2021. PMID 34035833
- [Derived] Horakova D, Boster A, Bertolotto A, Freedman MS, Firmino I, Cavalier SJ, Jacobs AK, Thangavelu K, Daizadeh N, Poole EM, Baker DP, Margolin DH, Ziemssen T; CARE-MS I, CARE-MS II, and CAMMS03409 Investigators. Proportion of alemtuzumab-treated patients converting from relapsing-remitting multiple sclerosis to secondary progressive multiple sclerosis over 6 years. Mult Scler J Exp Transl Clin. 2020 Dec 18;6(4):2055217320972137. doi: 10.1177/2055217320972137. eCollection 2020 Oct-Dec. PMID 33414927
- [Derived] Ziemssen T, Bass AD, Berkovich R, Comi G, Eichau S, Hobart J, Hunter SF, LaGanke C, Limmroth V, Pelletier D, Pozzilli C, Schippling S, Sousa L, Traboulsee A, Uitdehaag BMJ, Van Wijmeersch B, Choudhry Z, Daizadeh N, Singer BA; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ investigators. Efficacy and Safety of Alemtuzumab Through 9 Years of Follow-up in Patients with Highly Active Disease: Post Hoc Analysis of CARE-MS I and II Patients in the TOPAZ Extension Study. CNS Drugs. 2020 Sep;34(9):973-988. doi: 10.1007/s40263-020-00749-x. PMID 32710396
- [Derived] Gilmore W, Lund BT, Li P, Levy AM, Kelland EE, Akbari O, Groshen S, Cen SY, Pelletier D, Weiner LP, Javed A, Dunn JE, Traboulsee AL. Repopulation of T, B, and NK cells following alemtuzumab treatment in relapsing-remitting multiple sclerosis. J Neuroinflammation. 2020 Jun 15;17(1):189. doi: 10.1186/s12974-020-01847-9. PMID 32539719
- [Derived] Comi G, Alroughani R, Boster AL, Bass AD, Berkovich R, Fernandez O, Kim HJ, Limmroth V, Lycke J, Macdonell RA, Sharrack B, Singer BA, Vermersch P, Wiendl H, Ziemssen T, Jacobs A, Daizadeh N, Rodriguez CE, Traboulsee A; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ Investigators. Efficacy of alemtuzumab in relapsing-remitting MS patients who received additional courses after the initial two courses: Pooled analysis of the CARE-MS, extension, and TOPAZ studies. Mult Scler. 2020 Dec;26(14):1866-1876. doi: 10.1177/1352458519888610. Epub 2019 Nov 25. PMID 31762387
- [Derived] Van Wijmeersch B, Singer BA, Boster A, Broadley S, Fernandez O, Freedman MS, Izquierdo G, Lycke J, Pozzilli C, Sharrack B, Steingo B, Wiendl H, Wray S, Ziemssen T, Chung L, Margolin DH, Thangavelu K, Vermersch P. Efficacy of alemtuzumab over 6 years in relapsing-remitting multiple sclerosis patients who relapsed between courses 1 and 2: Post hoc analysis of the CARE-MS studies. Mult Scler. 2020 Nov;26(13):1719-1728. doi: 10.1177/1352458519881759. Epub 2019 Nov 1. PMID 31675266
- [Derived] Okai AF, Amezcua L, Berkovich RR, Chinea AR, Edwards KR, Steingo B, Walker A, Jacobs AK, Daizadeh N, Williams MJ; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ Investigators. Efficacy and Safety of Alemtuzumab in Patients of African Descent with Relapsing-Remitting Multiple Sclerosis: 8-Year Follow-up of CARE-MS I and II (TOPAZ Study). Neurol Ther. 2019 Dec;8(2):367-381. doi: 10.1007/s40120-019-00159-2. Epub 2019 Oct 25. PMID 31654272
- [Derived] Arroyo R, Bury DP, Guo JD, Margolin DH, Melanson M, Daizadeh N, Cella D. Impact of alemtuzumab on health-related quality of life over 6 years in CARE-MS II trial extension patients with relapsing-remitting multiple sclerosis. Mult Scler. 2020 Jul;26(8):955-963. doi: 10.1177/1352458519849796. Epub 2019 May 30. PMID 31144568
- [Derived] Li Z, Richards S, Surks HK, Jacobs A, Panzara MA. Clinical pharmacology of alemtuzumab, an anti-CD52 immunomodulator, in multiple sclerosis. Clin Exp Immunol. 2018 Dec;194(3):295-314. doi: 10.1111/cei.13208. Epub 2018 Oct 1. PMID 30144037
- [Derived] Arnold DL, Fisher E, Brinar VV, Cohen JA, Coles AJ, Giovannoni G, Hartung HP, Havrdova E, Selmaj KW, Stojanovic M, Weiner HL, Lake SL, Margolin DH, Thomas DR, Panzara MA, Compston DA; CARE-MS I and CARE-MS II Investigators. Superior MRI outcomes with alemtuzumab compared with subcutaneous interferon beta-1a in MS. Neurology. 2016 Oct 4;87(14):1464-1472. doi: 10.1212/WNL.0000000000003169. Epub 2016 Sep 2. PMID 27590291
- [Derived] Grafals M, Smith B, Murakami N, Trabucco A, Hamill K, Marangos E, Gilligan H, Pomfret EA, Pomposelli JJ, Simpson MA, Azzi J, Najafian N, Riella LV. Immunophenotyping and efficacy of low dose ATG in non-sensitized kidney recipients undergoing early steroid withdrawal: a randomized pilot study. PLoS One. 2014 Aug 11;9(8):e104408. doi: 10.1371/journal.pone.0104408. eCollection 2014. PMID 25111080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened at 192 investigational sites between October 10, 2007 and September 15, 2011.
Groups:
- Alemtuzumab 24mg: Alemtuzumab 24 mg per day IV infusion on 5 consecutive days at Month 0, followed by alemtuzumab 24 mg per day IV infusion on 3 consecutive days at Month 12.
Period: Overall Study
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg | Alemtuzumab 24mg
Started | 231 (Randomized.) | 436 (Randomized.) | 173 (Randomized.)
Treated | 202 (All randomized participants who received at least 1 dose of study drug as per initial randomization.) | 426 (All randomized participants who received at least 1 dose of study drug as per initial randomization.) | 170 (All randomized participants who received at least 1 dose of study drug as per initial randomization.)
Completed | 175 | 416 | 164
Not Completed | 56 | 20 | 9
Not completed — Adverse Event | 6 | 2 | 0
Not completed — Lack of Efficacy | 6 | 0 | 0
Not completed — Physician Decision | 3 | 4 | 1
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 36 | 12 | 5
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Death | 0 | 1 | 1
Not completed — Sponsor decision | 1 | 0 | 0
Not completed — Randomized but not treated | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population included all randomized participants who received at least 1 dose of study drug as per initial randomization.
Groups:
- Interferon Beta-1a: Interferon Beta-1a 44 mcg subcutaneously 3-times weekly for 24 months. Dose adjustment was done as per Investigator's discretion.
- Alemtuzumab 12 mg: Alemtuzumab 12 mg per day IV infusion on 5 consecutive days at Month 0, followed by alemtuzumab 12 mg per day IV infusion over 4 hours on 3 consecutive days at Month 12.
- Alemtuzumab 24mg: Alemtuzumab 24 mg per day IV infusion on 5 consecutive days at Month 0, followed by alemtuzumab 24 mg per day IV infusion over 4 hours on 3 consecutive days at Month 12.
- Total: Total of all reporting groups
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg | Alemtuzumab 24mg | Total
Number analyzed (Participants) | 202 | 426 | 170 | 798
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (8.77) | 34.8 (8.36) | 35.1 (8.40) | 35.1 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 281 | 120 | 532
  Male | 71 | 145 | 50 | 266
Time Since First Relapse [Median (Full Range); unit: years] | 4.1 [0.4 to 10.1] | 3.8 [0.2 to 14.4] | 3.7 [0.2 to 16.9] | 3.8 [0.2 to 16.9]
Number of Relapse Episodes in the Preceding 2 Years [Number; unit: participants] — Number of participants with 1, 2 or greater than or equal to 3 relapses are reported.
  participants
    1 Relapse | 7 | 15 | 11 | 33
    2 Relapses | 109 | 215 | 94 | 418
    Greater than or equal to 3 Relapses | 86 | 196 | 65 | 347
Expanded Disability Status Scale (EDSS) Score [Mean (Standard Deviation); unit: units on a scale] — EDSS is an ordinal scale in half-point increments that quantifies disability in participants with multiple sclerosis (MS). It assesses the 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS).
  units on a scale | 2.7 (1.21) | 2.7 (1.26) | 2.7 (1.17) | 2.7 (1.22)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Accumulation of Disability (SAD)
Description: EDSS is an ordinal scale in half-point increments that qualifies disability in participants with MS. It assesses 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score: 0 (normal neurological examination) to 10 (death due to MS). As measured by EDSS score, SAD was defined as increase of at least 1.5 points for participants with Baseline score of 0 and increase of at least 1.0 point for participants with a Baseline score of 1.0 or more; and the increase persisted for at least the next 2 scheduled assessments, that is, 6 consecutive months. The onset date of SAD was date of first EDSS assessment that began 6 month consecutive period of SAD. Participants who did not reach SAD endpoint were censored at their last visit. Percentage of participants with SAD, estimated by Kaplan-Meier (KM) method, was reported.
Time Frame: Up to 2 years
Population: FAS population included all randomized participants who received at least 1 dose of study drug as per initial randomization. Analysis was not performed for Alemtuzumab 24 mg as recruitment to this arm was closed early to reduce overall sample size, duration of enrollment period, overall duration of study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Alemtuzumab 12 mg: Alemtuzumab 12 mg per day IV infusion on 5 consecutive days at Month 0, followed by alemtuzumab 12 mg per day IV infusion on 3 consecutive days at Month 12.
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg
Number analyzed (Participants) | 202 | 426
percentage of participants | 21.13 [15.95 to 27.68] | 12.71 [9.89 to 16.27]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab 12 mg; Cox proportional hazards (PH) regression model with robust variance estimation using treatment group and geographic region as covariate was used; Test type: Superiority or Other; p = 0.0084, Cox Proportional Hazards Regression — Hochberg method was used to adjust for the two co-primary outcomes; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.38 to 0.87]

2. Primary Outcome: Annualized Relapse Rate
Description: Relapse was defined as new neurological symptoms or worsening of previous neurological symptoms with an objective change on neurological examination, attributable to multiple sclerosis that lasted for at least 48 hours, that were present at normal body temperature, and that were preceded by at least 30 days of clinical stability. Annualized relapse rate was estimated through negative binomial regression with robust variance estimation and covariate adjustment for geographic region using observed number of relapses as dependent variable, the log total amount of follow-up from date of first study treatment for each participant as an offset variable, and treatment group and geographic region as model covariates.
Time Frame: Up to 2 years
Population: FAS population. Analysis was not performed for Alemtuzumab 24 mg as described in outcome measure 1.
Measure: Number (95% Confidence Interval); unit: relapses per participant per year
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg
Number analyzed (Participants) | 202 | 426
relapses per participant per year | 0.52 [0.41 to 0.66] | 0.26 [0.21 to 0.33]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab 12 mg; Proportional means regression model with robust variance estimation and covariate adjustment for geographic region was used; Test type: Superiority or Other; p < 0.0001, Proportional means regression — Hochberg method was used to adjust for the two co-primary outcomes; Rate ratio = 0.51, 95% CI 2-sided [0.39 to 0.65]

3. Secondary Outcome: Percentage of Participants Who Were Relapse Free at Year 2
Description: Participants were considered relapse free at Year 2 if they did not experience a relapse from the date of first study treatment to study completion at 24 months. Percentage of participants who were relapse free at Year 2, estimated using the KM method, was reported.
Time Frame: Year 2
Population: FAS population. Analysis was not performed for Alemtuzumab 24 mg as described in outcome measure 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg
Number analyzed (Participants) | 202 | 426
percentage of participants | 46.70 [39.53 to 53.54] | 65.38 [60.65 to 69.70]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab 12 mg; Cox PH regression model with robust variance estimation and covariate adjustment for geographic region was used; Test type: Superiority or Other; p < 0.0001, Cox Proportional Hazards Regression; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.41 to 0.69]

4. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Score at Year 2
Description: EDSS is an ordinal scale in half-point increments that qualifies disability in participants with multiple sclerosis (MS). It assesses the 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS). Change was calculated by subtracting Baseline value from value at Year 2.
Time Frame: Baseline, Year 2
Population: FAS population. Here, number of participants analyzed was subset of FAS who had EDSS assessment at both Baseline and end-of-study (Year 2). Analysis was not performed for Alemtuzumab 24 mg as described in outcome measure 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg
Number analyzed (Participants) | 174 | 413
units on a scale | 0.21 (1.167) | -0.20 (1.084)
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab 12 mg; The analysis was performed using Wei-Lachin method for non-parametric analysis of repeated measures; Test type: Superiority or Other; p < 0.0001, Wei-Lachin

5. Secondary Outcome: Change From Baseline in Multiple Sclerosis Functional Composite (MSFC) Score at Year 2
Description: MSFC is a multidimensional measure consisting of quantitative tests of ambulation (Timed 25-Foot Walk), manual dexterity (9-Hole Peg Test; 9HPT), and cognitive function (Paced Auditory Serial Addition Test; PASAT). The MSFC score was calculated as the mean of the Z-scores of the 3 components. A Z-score was calculated by subtracting the mean of the reference population from the test result, then dividing by the standard deviation of the reference population. Higher Z-scores reflected better neurological function and a positive change from Baseline indicates improvement. An increase in score indicated an improvement (Z-score range: -3 to +3). Acquisition of disability was measured by change from Baseline in MSFC score at Year 2.
Time Frame: Baseline, Year 2
Population: FAS population. Here, number of participants analyzed signifies subset of FAS who had MSFC score assessment at Baseline; 'n' signifies participants who had MSFC score assessment at Baseline (for Baseline) and at both Baseline and Year 2 (for change at Year 2). Analysis was not performed for Alemtuzumab 24 mg as described in outcome measure 1.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg
Number analyzed (Participants) | 198 | 423
Z-score
  Baseline (n=198, 423) | -0.03 (0.791) | 0.02 (0.689)
  Change at Year 2 (n=169, 399) | -0.04 (0.449) | 0.09 (0.358)
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab 12 mg; Change at Year 2: the analysis was performed using Wei-Lachin method for non-parametric analysis of repeated measures; Test type: Superiority or Other; p = 0.0022, Wei-Lachin

6. Secondary Outcome: Percent Change From Baseline in Magnetic Resonance Imaging Time Constant 2 (MRI-T2) Hyperintense Lesion Volume at Year 2
Description: Percent change in MS lesion volume as measured by MRI-T2 scan was calculated from MRI-T2-weighted scans as the following: (lesion volume at 2 years - lesion volume at Baseline)*100/ (lesion volume at Baseline).
Time Frame: Baseline, Year 2
Population: FAS population. Here, number of participants analyzed was subset of FAS who had assessment for T2 volume at both Baseline and end-of-study (Year 2). Analysis was not performed for Alemtuzumab 24 mg as described in outcome measure 1.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg
Number analyzed (Participants) | 190 | 412
percent change | 2.41 (26.48) | -1.12 (24.40)
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab 12 mg; Ranked ANCOVA models with covariate adjustment for geographic region and Baseline T2 lesion volume was used; Test type: Superiority or Other; p = 0.1371, Ranked ANCOVA

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 2 years
Description: If a participant experienced a serious and a non-serious event with same term, individual was included in numerator of both adverse event tables. Safety population: all participants who received any amount of study drug (as treated). In Alemtuzumab 24 mg arm 9 participants received Alemtuzumab 12 mg, hence were included in Alemtuzumab 12 mg arm.
Groups:
- Alemtuzumab (Pooled): Included all participants who received alemtuzumab 12 mg or 24 mg per day IV infusion on 5 consecutive days at Month 0, followed by alemtuzumab 12 mg or 24 mg per day IV infusion on 3 consecutive days at Month 12.
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg | Alemtuzumab 24 mg | Alemtuzumab (Pooled)
Serious Adverse Events (participants affected / at risk) | 44/202 | 85/435 | 30/161 | 115/596
Other Adverse Events (participants affected / at risk) | 189/202 | 427/435 | 159/161 | 586/596
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Beta-1a (N=202) | Alemtuzumab 12 mg (N=435) | Alemtuzumab 24 mg (N=161) | Alemtuzumab (Pooled) (N=596)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2 | 1 | 3
Eye pain (Eye disorders) | 0 | 1 | 0 | 1
Retinal pigment epitheliopathy (Eye disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Sigmoiditis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Abasia (General disorders) | 0 | 0 | 1 | 1
Chest discomfort (General disorders) | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 2 | 0 | 2
Death (General disorders) | 0 | 1 | 0 | 1
Infusion related reaction (General disorders) | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 2
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 2 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2 | 0 | 2
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 1 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 2 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Catheter site infection (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 1
Febrile infection (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 3 | 1 | 4
Herpes zoster (Infections and infestations) | 0 | 1 | 2 | 3
Influenza (Infections and infestations) | 0 | 1 | 0 | 1
Injection site abscess (Infections and infestations) | 1 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 1 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 1
Pasteurella infection (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 4 | 1 | 5
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 1
Intracranial hypotension (Nervous system disorders) | 0 | 1 | 1 | 2
Migraine (Nervous system disorders) | 0 | 1 | 1 | 2
Monoparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1 | 1
Multiple sclerosis relapse (Nervous system disorders) | 25 | 33 | 3 | 36
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 1 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 1
Status migrainosus (Nervous system disorders) | 0 | 1 | 0 | 1
Drug dependence (Psychiatric disorders) | 0 | 1 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Mania (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1 | 2
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 1
Automatic bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 1 | 2
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vulvar dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3
Female sterilisation (Surgical and medical procedures) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Beta-1a (N=202) | Alemtuzumab 12 mg (N=435) | Alemtuzumab 24 mg (N=161) | Alemtuzumab (Pooled) (N=596)
Lymphopenia (Blood and lymphatic system disorders) | 4 | 23 | 9 | 32
Tachycardia (Cardiac disorders) | 1 | 27 | 10 | 37
Vision blurred (Eye disorders) | 10 | 21 | 9 | 30
Abdominal pain (Gastrointestinal disorders) | 6 | 23 | 18 | 41
Abdominal pain upper (Gastrointestinal disorders) | 6 | 16 | 11 | 27
Constipation (Gastrointestinal disorders) | 15 | 19 | 14 | 33
Diarrhoea (Gastrointestinal disorders) | 17 | 58 | 34 | 92
Dyspepsia (Gastrointestinal disorders) | 9 | 32 | 19 | 51
Nausea (Gastrointestinal disorders) | 21 | 105 | 51 | 156
Vomiting (Gastrointestinal disorders) | 8 | 39 | 26 | 65
Asthenia (General disorders) | 10 | 22 | 9 | 31
Chest discomfort (General disorders) | 1 | 32 | 27 | 59
Chills (General disorders) | 9 | 35 | 22 | 57
Fatigue (General disorders) | 26 | 81 | 35 | 116
Influenza like illness (General disorders) | 47 | 31 | 13 | 44
Injection site erythema (General disorders) | 28 | 0 | 0 | 0
Injection site reaction (General disorders) | 13 | 0 | 0 | 0
Oedema peripheral (General disorders) | 4 | 26 | 12 | 38
Pain (General disorders) | 7 | 35 | 16 | 51
Pyrexia (General disorders) | 18 | 94 | 47 | 141
Bronchitis (Infections and infestations) | 10 | 34 | 15 | 49
Gastroenteritis (Infections and infestations) | 5 | 20 | 9 | 29
Gastroenteritis viral (Infections and infestations) | 12 | 17 | 8 | 25
Herpes zoster (Infections and infestations) | 3 | 24 | 12 | 36
Influenza (Infections and infestations) | 11 | 40 | 18 | 58
Nasopharyngitis (Infections and infestations) | 48 | 128 | 52 | 180
Oral herpes (Infections and infestations) | 4 | 35 | 9 | 44
Pharyngitis (Infections and infestations) | 1 | 19 | 9 | 28
Sinusitis (Infections and infestations) | 20 | 58 | 20 | 78
Upper respiratory tract infection (Infections and infestations) | 25 | 70 | 34 | 104
Urinary tract infection (Infections and infestations) | 23 | 92 | 37 | 129
Contusion (Injury, poisoning and procedural complications) | 15 | 50 | 30 | 80
Fall (Injury, poisoning and procedural complications) | 11 | 28 | 10 | 38
Bacterial test positive (Investigations) | 4 | 13 | 9 | 22
CD4 lymphocytes decreased (Investigations) | 2 | 23 | 9 | 32
CD8 lymphocytes decreased (Investigations) | 4 | 23 | 7 | 30
Lymphocyte count decreased (Investigations) | 5 | 18 | 11 | 29
Platelet count decreased (Investigations) | 12 | 16 | 1 | 17
T-lymphocyte count decreased (Investigations) | 5 | 16 | 10 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 57 | 26 | 83
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 52 | 30 | 82
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 28 | 12 | 40
Muscular weakness (Musculoskeletal and connective tissue disorders) | 14 | 29 | 15 | 44
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 34 | 24 | 58
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 65 | 26 | 91
Dizziness (Nervous system disorders) | 11 | 48 | 26 | 74
Dysgeusia (Nervous system disorders) | 8 | 29 | 14 | 43
Headache (Nervous system disorders) | 35 | 230 | 101 | 331
Hypoaesthesia (Nervous system disorders) | 16 | 35 | 19 | 54
Migraine (Nervous system disorders) | 11 | 11 | 6 | 17
Multiple sclerosis relapse (Nervous system disorders) | 84 | 119 | 51 | 170
Paraesthesia (Nervous system disorders) | 20 | 50 | 18 | 68
Tremor (Nervous system disorders) | 3 | 14 | 10 | 24
Anxiety (Psychiatric disorders) | 14 | 31 | 16 | 47
Depression (Psychiatric disorders) | 25 | 29 | 16 | 45
Insomnia (Psychiatric disorders) | 28 | 69 | 32 | 101
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 35 | 22 | 57
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 37 | 27 | 64
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 23 | 7 | 30
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 47 | 24 | 71
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 9 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 12 | 10 | 22
Erythema (Skin and subcutaneous tissue disorders) | 3 | 23 | 12 | 35
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 66 | 35 | 101
Rash (Skin and subcutaneous tissue disorders) | 11 | 193 | 95 | 288
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 33 | 16 | 49
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 9 | 11 | 20
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 74 | 42 | 116
Flushing (Vascular disorders) | 7 | 34 | 16 | 50

LIMITATIONS AND CAVEATS:
Efficacy analysis was not performed for Alemtuzumab 24 mg as recruitment to this arm was closed early to reduce overall sample size, duration of enrollment period, overall duration of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can publish after sponsor published, after a defined period of time after study completion, and/or with written Sponsor approval. Generally PI gives sponsor a draft 60 days before publication. Sponsor can ask that confidential information can be removed, and can further defer publication upon notifying PI that it will file a patent application on inventions contained in the draft.